CLINICAL TRIAL: NCT01241578
Title: Improving Behavioral Weight Loss Via Electronic Handheld Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Principal Investigator, John Graham Thomas, Assistant Professor (Research), The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOSNewInvestigator2009
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Obesity; Behavior Therapy; Lifestyle; Technology; Cellular Phone
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile Phone Intervention (Experimental): Participants receive a behavioral intervention via mobile phone and brief in-person counseling sessions.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Participants receive instructions for making healthy changes to their diet and physical activity habits.

SUMMARY:
Standard behavioral treatment (SBT) for obesity is often effective, but weight losses are highly variable, and patients sometimes fail to achieve a "successful" weight loss of 5-10% of their starting weight. It has been suggested that the "one size fits all" approach of SBT may be responsible for many treatment failures because the intervention is not sufficiently tailored to address the unique needs of each patient. Moreover, treatment is delivered in the clinic, not in the settings and the times when it is needed most. The primary aim of the proposed research is to develop and pilot test a behavioral weight loss intervention that combines in-person sessions with treatment delivered via an electronic handheld device to provide highly individualized weight loss treatment in patients' natural environment. In a critical departure from previous research using cell phone technology, the portion of intervention that is delivered via handheld device will be of equal sophistication and importance to the portion of the intervention that is delivered in face-to-face treatment sessions. The proposed study seeks to determine the feasibility and preliminary efficacy of an individually tailored behavioral weight loss program that integrates clinic-based care and smartphone technology.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (kg/m2) of 30-45.
* English language fluency
* Basic familiarity with cell phone technology
* Ability to read at a 6th grade level
* Availability to attend weekly treatment sessions in Providence, RI

Exclusion Criteria:

* Any heart condition that limits ability to participate in physical activity
* Chest Pain
* Any cognitive of physical limitation that would preclude use of a smartphone
* Serious mental illness
* Historical or current eating disorder
* Previous or planned bariatric surgery
* Use of weight loss medication
* Recent pregnancy or a plan to become pregnant in the next 6 months
* Participation in a study at the Weight Control and Diabetes Research Center within the last two years
* A weight loss of greater than 5% body weight in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline and weekly for 24-weeks.
  Participants' body weight measured in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thomas, Ph.D., Principal Investigator — Brown University; Rena R Wing, Ph.D., Principal Investigator — Brown University
Locations (1):
- Weight Control and Diabetes Resarch Center, Providence, Rhode Island, United States